CLINICAL TRIAL: NCT02152644
Title: Prevalence of Amyloidosis in Carpal Tunnel Surgery
Brief Title: Prevalence of Amyloidosis and Carpal Tunnel
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1589
Record Dates: First submitted 2014-04-01; First posted 2014-06-02 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Amyloid Neuropathy, Carpal Tunnel
Keywords: amyloidosis-carpal tunnel
MeSH Terms: conditions — Amyloid Neuropathies; Median Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- amyloid: unique cohort of Adult patients older than 21 years with carpal tunnel syndrome with surgical indication (moderate to severe symptoms that do not respond to conservative treatment physiotherapy, splinting, activity modification) for more than 6 months.

SUMMARY:
This is a cross sectional study to estimate the prevalence of the presence of amyloid deposits in a biopsy of subcutaneous fat cell, carpal flexor retinaculum and synovial tissue sheath of the flexor tendons requirement for carpal tunnel surgery.

DETAILED DESCRIPTION:
Amyloidosis (A) is a disease caused by the deposit of usually misfolded protein in form of amorphous fibrillar material in different tissues, which may cause their progressive dysfunction. The prevalence of amyloidosis varies by population studied and the type of amyloid. Although the prevalence in the general population is unknown, the Mayo Clinic in U.S. estimated a 1/90666. This disease generated about 0.0084 % (1367/16232579) of total hospital visits between April 2008 and April 2009 in England.

The most frequent clinical manifestations are cardiac, renal and hepatic involvement, but vary widely depending on the type of amyloidosis , organ affected and the extent of the deposits. Infiltration of amyloid may produce signs and symptoms that could be very similar to other diseases, like the rheumatologic one. This potentially polymorphous clinic presentation may suggest under-diagnosis by low clinical suspicion.

Carpal tunnel syndrome is frequent in patients with A and may be the initial manifestation. This syndrome is generated by the progressive infiltration of amyloid fibrils in the retinaculum flexor and in synovial tissue, causing compression of the medium nerve. A frequency of up to 13% of carpal tunnel syndrome has been reported in patients with primary amyloidosis.

In 1993, Breda et al. assessed 98 tendon and synovial tissue's biopsies of patients operated for carpal tunnel syndrome. The pathology revealed amyloid deposition in 12% of them, of which 8 had no evidence of systemic disease. This amyloid deposition was interpreted as probably secondary to chronic local inflammation. In 1992, Kyle et al. evaluated the incidence of systemic amyloidosis in a retrospective cohort of 35 patients with carpal tunnel syndrome and synovial local deposition of amyloidosis without evidence of systemic amyloidosis. During follow-up only 2 developed systemic amyloidosis and 11 showed only laboratory abnormalities (9 monoclonal band and 2 monoclonal light chain in the urine). In this group the amyloid deposition was identified as transthyretin (TTR) dependent in 32 of 35 cases.

Even though there are estimations regarding the prevalence of A in general populations worldwide and in patients with carpal tunnel syndrome surgery, there is no local estimation in Argentina. Additionally, it is not known if the presentation of amyloid deposits in tendon elements of pathological the carpal tunnel correlates with subcutaneous amyloid deposit.

In this project the investigators propose to estimate the prevalence of Amyloidosis in the synovial tissue of patients with surgical carpal tunnel syndrome and correlate them with deposits of amyloid in the subcutaneous cellular tissue fat.

What is the prevalence of amyloidosis, in cellular subcutaneous fat biopsy, flexor retinaculum of the carpus and synovial tissue of the flexor tendons sheath, in patients with carpal tunnel syndrome surgery?

Primary objective

1. To estimate the prevalence of the presence of amyloid deposits in: (i) a biopsy of cellular subcutaneous fat, (ii) the flexor retinaculum of the carpus and (iii) synovial tissue of the flexor tendons sheath, with requirement for carpal tunnel surgery.

Secondary objectives

1. Detect and characterize patients with subclinical amyloidosis.
2. Identify the protein deposited in patients with amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 21 years with carpal tunnel syndrome with surgical indication (moderate to severe symptoms that do not respond to conservative treatment physiotherapy, splinting, activity modification) for more than 6 months.

Exclusion Criteria:

* Refusal to participate or to the process of informed consent.
* Secondary acute carpal tunnel syndrome (eg ganglion).
* Formal contraindication surgical treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients older than 21 years with carpal tunnel syndrome with surgical indication (moderate to severe symptoms that do not respond to conservative treatment physiotherapy, splinting, activity modification) for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
presence of amyloid deposits | one month

CONTACTS AND LOCATIONS:
Overall Officials: Adela Aguirre, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Lourdes Posadas-Martínez, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Dorotea Fantl, MD, Principal Investigator — Hospital Italiano de Buenos Aires; María S. Saez, BCH, Principal Investigator — Hospital Italiano de Buenos Aires; Gustavo Greloni, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Federico Varela, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Patricia Sorroche, BCH, Principal Investigator — Hospital Italiano de Buenos Aires; Gabriel Waisman, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Fernán G. De Quiros, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Jorge Boretto, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Elsa Nucifora, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Diego Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- HIBA, CABA, Buenos Aires, Argentina